CLINICAL TRIAL: NCT02288091
Title: A Pilot Study of Inosine in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Salah Foundation (Other); Sean M. Healey & AMG Center for ALS (Other)
Responsible Party: Principal Investigator, Sabrina Paganoni, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 701
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Inosine; Uric acid; Urate; Glutathione; Biomarker; Oxidative stress; Oxidative damage; proof-of-concept
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Inosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label (Experimental): Subjects will receive oral inosine daily.
  Interventions: Drug: Inosine

INTERVENTIONS:
Drug: Inosine — Twenty-five eligible subjects will receive inosine for 12 weeks (administered in the form of 500 mg capsules, 1 to 6 capsules a day for a total daily dose of up to 3 gm). The dose of inosine will be titrated to target urate levels of 7-8 mg/dL based on urate level measurement that will occur at Week 2, Week 4, Week 6, and Week 9 after Baseline.

SUMMARY:
This is a single center, open label, 12-week study of inosine treatment. Inosine treatment leads to an increase in the levels of urate (uric acid) in the blood.

The primary objective of the study is to determine the tolerability of oral administration of inosine.

Secondary study objectives include the measurement of biomarkers of oxidative stress and damage in response to inosine treatment.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal, neurodegenerative disease for which there is no cure. Multiple lines of evidence have implicated oxidative stress in the pathophysiology of ALS. Urate (uric acid) is an endogenous antioxidant system, and urate may serve as a major defense against oxidative stress. Urate has emerged as a promising neuro-protectant and therapeutic target based on convergent epidemiological, laboratory, and clinical data in multiple neurodegenerative diseases, most notably Parkinson's disease (PD). In PD, urate elevation has been pursued as a potential therapy by administration of inosine, a urate precursor that is available as an over-the-counter supplement. Administration of inosine results in a predictable elevation of urate levels and has been shown to be safe and well tolerated in PD.

Analysis of ALS databases revealed that higher urate levels are an independent predictor of slower progression and prolonged survival in ALS. However, whether elevating urate in people with ALS would result in better outcomes is unknown. As a first step towards development of inosine as a potential treatment for ALS, in this study we will test whether inosine administration in ALS is safe and correlates with changes in the levels of biomarkers of oxidative stress and damage (as biomarkers of the intended biological effect).

The primary outcome measures will be safety, as measured by adverse events and clinically meaningful changes in vital signs, physical examination, and standard clinical laboratory tests, and tolerability, defined as the ability of subjects to complete the entire 12-week study.

The secondary objective of the study is to quantify the effect of the treatment on biomarkers of oxidative damage and stress.

An exploratory objective of the study is to measure whether changes in these biomarkers are different in people with bulbar-onset ALS compared to people with limb-onset ALS.

This study will be conducted in people who meet the El Escorial criteria of possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS. At screening, eligible individuals must be at least 18 years old and must provide written informed consent prior to screening. Subjects on a stable dose of riluzole and those not taking riluzole, and women of child-bearing age at screening are eligible for inclusion as long as they meet specific protocol requirements.

Study participants will be administered oral inosine daily. The dose of inosine will be titrated to obtain serum urate levels of 7 - 8 mg/dL.

Study participants will remain on treatment until the Week 12 visit. Each participant will also have a Week 16 Follow-up Telephone Interview to assess for adverse events (AEs), changes in concomitant medications and to administer the ALSFRS-R.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria (Appendix 1).
3. Capable of providing informed consent and following trial procedures.
4. Serum urate < 5.5 mg/dl at screening (i.e. below the population median serum urate levels).
5. Willingness to undergo magnetic resonance spectroscopy (MRS) at Baseline and at Week 12 of the study.
6. Women must not be able to become pregnant (e.g. post menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and 3 months after study completion. Adequate contraception includes: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal (patch or contraceptive ring, for example) contraception), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.

Exclusion Criteria:

1. History of urolithiasis.
2. Urine pH < 5.5 at screening (as acidic urine is a major determinant of uric acid urolithiasis).
3. Urate crystalluria at Screening.
4. History of gout.
5. History of stroke or myocardial infarction.
6. History of symptomatic coronary artery disease (e.g. angina pectoris) or symptomatic peripheral arterial disease within 1 year prior to Screening.
7. Symptomatic congestive heart failure with a documented ejection fraction below 45%.
8. Poorly controlled arterial hypertension (SBP>160mmHg or DBP>100mmHg at Screening).
9. Contraindications to undergo magnetic resonance spectroscopy (MRS) at Baseline and at Week 12 of the study such as history of claustrophobia, inability to lie flat for approximately one hour, or metal implants (metal pins or plates, extensive non-removable dental work, cerebral aneurysm clips, pacemaker).
10. Women who are pregnant or lactating.
11. The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, according to PI judgment, or a history of active substance abuse within the prior year.
12. Anything that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
13. Use of the following within 30 days prior to Screening: inosine, allopurinol, probenecid, more than 300mg vitamin C daily (note that a subject may take a standard multivitamin up to one tablet or capsule daily). Use of thiazides is permissible as long as the subject is on a stable dose from 1 week prior to Screening.
14. Known hypersensitivity or intolerability to inosine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Paganoni, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paganoni S, Zhang M, Quiroz Zarate A, Jaffa M, Yu H, Cudkowicz ME, Wills AM. Uric acid levels predict survival in men with amyotrophic lateral sclerosis. J Neurol. 2012 Sep;259(9):1923-8. doi: 10.1007/s00415-012-6440-7. Epub 2012 Feb 10. PMID 22323210
- [Background] Atassi N, Berry J, Shui A, Zach N, Sherman A, Sinani E, Walker J, Katsovskiy I, Schoenfeld D, Cudkowicz M, Leitner M. The PRO-ACT database: design, initial analyses, and predictive features. Neurology. 2014 Nov 4;83(19):1719-25. doi: 10.1212/WNL.0000000000000951. Epub 2014 Oct 8. PMID 25298304
- [Background] Parkinson Study Group SURE-PD Investigators; Schwarzschild MA, Ascherio A, Beal MF, Cudkowicz ME, Curhan GC, Hare JM, Hooper DC, Kieburtz KD, Macklin EA, Oakes D, Rudolph A, Shoulson I, Tennis MK, Espay AJ, Gartner M, Hung A, Bwala G, Lenehan R, Encarnacion E, Ainslie M, Castillo R, Togasaki D, Barles G, Friedman JH, Niles L, Carter JH, Murray M, Goetz CG, Jaglin J, Ahmed A, Russell DS, Cotto C, Goudreau JL, Russell D, Parashos SA, Ede P, Saint-Hilaire MH, Thomas CA, James R, Stacy MA, Johnson J, Gauger L, Antonelle de Marcaida J, Thurlow S, Isaacson SH, Carvajal L, Rao J, Cook M, Hope-Porche C, McClurg L, Grasso DL, Logan R, Orme C, Ross T, Brocht AF, Constantinescu R, Sharma S, Venuto C, Weber J, Eaton K. Inosine to increase serum and cerebrospinal fluid urate in Parkinson disease: a randomized clinical trial. JAMA Neurol. 2014 Feb;71(2):141-50. doi: 10.1001/jamaneurol.2013.5528. PMID 24366103

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label
Started | 32
Randomized/Treated | 25
Completed | 24
Not Completed | 8
Not completed — Lost to Follow-up | 1
Not completed — Screen fail | 7

BASELINE CHARACTERISTICS:
Population: 32 subjects were consented, however, 25 patients were randomized/treated to received the study drug.
Arm/Group | Open-label
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 32 subjects were consented, however, 25 patients were randomized/treated to received the study drug.
  Participants
    Female | 18
    Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 32 subjects were consented, however, 25 patients were randomized/treated to received the study drug.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 24
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 32 subjects were consented, however, 25 patients were randomized/treated to received the study drug.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 23
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: 32 subjects were consented, however, 25 patients were randomized/treated to received the study drug.
  participants
    United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Safety will be assessed by the occurrence of adverse events.
Time Frame: 12 weeks
Population: No expected adverse events of special interest, such as kidney stones and gout, occurred during the course of the study. However, twenty-two (22) out of twenty-five (25) participants did experience an adverse event during the course of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label
Number analyzed (Participants) | 25
Participants | 22

2. Primary Outcome: Tolerability to Complete the Entire 12 Week Study on Study Drug.
Description: Tolerability will be defined as the ability of subjects to complete the entire 12-week study on study drug.
Time Frame: 12 weeks
Population: Twenty-four (24) out of twenty-five (25) participants completed 12 weeks of study drug treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label
Number analyzed (Participants) | 25
Participants | 24

3. Secondary Outcome: Blood Biomarkers (GSH) at Baseline and Week 12
Description: Blood samples will be obtained at baseline and after 12 weeks of treatment to measure biomarkers of oxidative stress and damage such as glutathione (GSH).
Time Frame: 12 weeks
Population: Two (2) subjects did not have blood drawn for GSH analysis at the Baseline Visit. Five (5) subjects did not have blood drawn for GSH analysis at the Week 12 visit. These missing samples are due to technical issues, such as a difficult blood draw or issue with sample processing.
Measure: Mean (Standard Deviation); unit: ƥM
Arm/Group | Open-label
Number analyzed (Participants) | 23
ƥM
  Glutathione at Baseline | 94.0 (28.4)
  Glutathione at Week 12: number analyzed (Participants) | 20
  Glutathione at Week 12 | 84.5 (42.6)

4. Secondary Outcome: Neuroimaging Biomarkers at Baseline and Week 12
Description: Magnetic resonance spectroscopy (MRS) will be performed to measure the levels of glutathione in the motor cortex; levels of glutathione at Week 12 (post-treatment) will be compared to pre-treatment levels.
Time Frame: 12 weeks
Population: Five (5) subjects did not have a MRS done at the Baseline and Week 12 visits. Of the 20 that had a baseline MRS, 2 patients did not have a Week 12 MRS done. These missing MRS scans are due to technical difficulties, such as subjects were unable to complete the scan.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Open-label
Number analyzed (Participants) | 20
mM
  Motor Cortex Precentral Gyri (Baseline) | 0.424 (0.064)
  Motor Cortex Precentral Gyri (Week 12): number analyzed (Participants) | 18
  Motor Cortex Precentral Gyri (Week 12) | 0.392 (0.064)

5. Secondary Outcome: Blood Biomarkers (FRAP) at Baseline and Week 12
Description: Blood samples will be obtained at baseline and after 12 weeks of treatment to measure biomarkers of oxidative stress and damage such as ferric reducing antioxidant power (FRAP).
Time Frame: 12 weeks
Population: One (1) subject did not have blood drawn for FRAP analysis at the Baseline Visit. Four (4) subjects did not have blood drawn for FRAP analysis at the Week 12 visit. These missing samples are due to technical issues, such as a difficult blood draw or issue with sample processing.
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Open-label
Number analyzed (Participants) | 24
µM
  Ferric Reducing Antioxidant Power (Baseline) | 765.7 (155.1)
  Ferric Reducing Antioxidant Power (Week 12): number analyzed (Participants) | 21
  Ferric Reducing Antioxidant Power (Week 12) | 1188.3 (294.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent until 28 days after a subject's last dose of study drug.
Arm/Group | Open-label
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (N=25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (N=25)
Weight Loss (Investigations) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Dysphagia aggravated (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Weakness worsened (General disorders) | 3 (3)
Ankle sprain (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Weakness of arms (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes